CLINICAL TRIAL: NCT06730191
Title: Free Buccal Pad Graft Versus Free Palatal Gingival Tissue Graft for Primary Soft Tissue Closure Over Immediately Placed Dental Implant in Maxillary Molar Socket
Brief Title: Soft Tissue Graft Over Immediately Placed Dental Implant in Maxillary Molar Socket
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Mai Ahmed Haggag (Other)
Responsible Party: Sponsor-Investigator, Mai Ahmed Haggag, Associate professor of oral and maxillofacial surgery, Mansoura University
Organization: Mansoura University (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: M01050230S
Record Dates: First submitted 2024-12-08; First posted 2024-12-12 (Actual); Last update posted 2024-12-12 (Actual); Status verified 2024-09

CONDITIONS: Dental Diseases
MeSH Terms: conditions — Stomatognathic Diseases

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- conventional (Other): conventional without anything only immediate dental implant covering by soft tissue graft
  Interventions: Procedure: soft tissue graft covering immediate dental implant
- Split thickness (Other): split thickness graft before covering immediate implant
  Interventions: Procedure: soft tissue graft covering immediate dental implant

INTERVENTIONS:
Procedure: soft tissue graft covering immediate dental implant — soft tissue graft covering immediate dental implant

SUMMARY:
Compare between free tissue graft of buccal pad of fat BFP and free palatal gingival tissue graft for primary soft tissue closure over immediately placed dental implant

DETAILED DESCRIPTION:
Buccal pad of fat BFP and free palatal gingival tissue graft over immediately placed dental implant

ELIGIBILITY:
Inclusion Criteria:

* class one molar extraction socket

Exclusion Criteria:

* pregnant females psychiatric problems

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 2 (Estimated)
Dates: Start 2025-07-11 (Estimated); Primary Completion 2025-12-11 (Estimated); Study Completion 2026-07-11 (Estimated)

PRIMARY OUTCOMES:
Soft tissue healing | 1,2,3,4,weeks
  Soft tissue healing by photograph

CONTACTS AND LOCATIONS:
Overall Officials: mansoura university, Principal Investigator — Mansoura University

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Rajan SA, Ramabhadran BK, Emmatty R, Paul TP, Jose P, Ameyaroy DK, Variath PT, Joseph M. Comparative Evaluation of Different Soft Tissue Coverage Techniques at Immediate Implant Sites: A Cohort Study. J Contemp Dent Pract. 2021 Nov 1;22(11):1268-1274. PMID 35343452
- [Background] Bleyan S, Gaspar J, Huwais S, Schwimer C, Mazor Z, Mendes JJ, Neiva R. Molar Septum Expansion with Osseodensification for Immediate Implant Placement, Retrospective Multicenter Study with Up-to-5-Year Follow-Up, Introducing a New Molar Socket Classification. J Funct Biomater. 2021 Nov 25;12(4):66. doi: 10.3390/jfb12040066. PMID 34940545